CLINICAL TRIAL: NCT02329106
Title: Comparison Percutaneous Cryosurgery and Irreversible Electroportion in Unresectable Liver Cancer Close to Diaphragmatic Dome
Brief Title: Percutaneous Irreversible Electroportion in Unresectable Liver Cancer Close to Diaphragmatic Dome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JF-20141225
Record Dates: First submitted 2014-12-26; First posted 2014-12-31 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2019-05

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Electroporation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NanoKnife LEDC System (Experimental): Ablation with the NanoKnife Low Energy Direct Current (LEDC) System, alao called Irreversible electroporation (IRE), 90 pulses of 70 microseconds each in duration will be administered per electrode pair.
  Interventions: Device: Irreversible electroporation (IRE)
- Control (No Intervention): The patients without treatment

INTERVENTIONS:
Device: Irreversible electroporation (IRE) — Irreversible electroporation (IRE) is a new, minimal-invasive image-guided treatment method for tumors not amenable for surgical resection or thermal ablation, due to vicinity near vital structures such as vessels,bile ducts and diaphragmatic dome.
  Other Names: NanoKnife
  Arms: NanoKnife LEDC System

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of irreversible electroportion in unresectable liver cancer close to diaphragmatic dome.

DETAILED DESCRIPTION:
Single-arm pilot clinical trial. Patients will be subjected to irreversible electroporation (IRE) as the sole treatment of liver cancer close to diaphragmatic dome.

This pilot study was designed to study the feasibility and safety of treatment as an alternative therapeutic IRE in the treatment of neoplastic nodules in the liver, with particular reference to close to diaphragmatic dome, where the current therapeutic arsenal is inadequate or counter-indicated.

To perform the IRE procedure the IRE NanoKnife™ System (AngioDynamics) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Liver cancer diagnosed by positive biopsy or non-invasive criteria,
* Tumors from diaphragm is <1 cm
* not suitable for surgical resection or transplantation,
* have at least one, but less than or equal to 3 tumors,
* of the tumour(s) identified, each tumor must be ≤ 5 cm in diameter,
* Child-Pugh class A,B
* Eastern Cooperative Oncology Group (ECOG) score of 0-1,
* a prothrombin time ratio > 50%,
* platelet count > 80x109/L,
* ability of patient to stop anticoagulant and anti-platelet therapy for seven days prior to and seven days post NanoKnife procedure,
* are able to comprehend and willing to sign the written informed consent form (ICF),
* have a life expectancy of at least 3 months.

Exclusion Criteria:

* liver cancer developed on an already transplanted liver,
* cardiac insufficiency, ongoing coronary artery disease or arrhythmia,
* any active implanted device (eg Pacemaker),
* women who are pregnant or women of child-bearing potential who are not using an acceptable method of contraception,
* have received treatment with an investigational agent/ procedure within 30 days prior to treatment with the NanoKnife™ LEDC System,
* are in the opinion of the Investigator unable to comply with the visit schedule and protocol evaluations.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of IRE for unresectable liver cancer close to diaphragmatic dome using Common terminology Criteria for Adverse Events (CTCAE). | up to 7 days
  Safety using Common terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Evaluate the efficacy of IRE for unresectable liver cancer close to diaphragmatic as measured by cell death of CRLM after IRE is demonstrated macroscopically by using vitality-staining with triphenyl-tetrazoliumchloride (TTC) | 1 year
  Cell death of CRLM after IRE is demonstrated macroscopically by using vitality-staining with triphenyl-tetrazoliumchloride (TTC). Since and shape of the ablation zone is assessed. Immunohistologic examination is used to more specifically assess microscopic cell damage and vessel wall damage. Apoptotic markers are used.

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi Niu, M.D.,PHD., Study Chair — President
Locations (1):
- FUDA Cancer Hospital, Guangzhou, Guangdong, China